CLINICAL TRIAL: NCT04732286
Title: A Phase IIIb, Single Arm, Multicenter Study of Atezolizumab in Combination With Bevacizumab to Investigate Safety and Efficacy in Spanish Patients With Unresectable or Unsuitable for Locoregional Treatments Hepatocellular Carcinoma Not Previously Treated With Systemic Therapy
Brief Title: A Study of Atezolizumab in Combination With Bevacizumab in Spanish Patients With Unresectable or Unsuitable for Locoregional Treatments Hepatocellular Carcinoma Not Previously Treated With Systemic Therapy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was completed as pre-specified in the protocol. Study was terminated only for participants who were in the study even after 24 months of follow-up as specified in the protocol.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML42600
Record Dates: First submitted 2021-01-28; First posted 2021-02-01 (Actual); Results first posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — atezolizumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm A (atezolizumab plus bevacizumab) (Experimental): Participants will receive Atezolizumab + Bevacizumab until unacceptable toxicity or loss of clinical benefit as determined by the investigator.
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab will be administered intravenously at a dose of 1200 mg on Day 1 of each 21-day cycle.
  Other Names: Tecentriq
Drug: Bevacizumab — Bevacizumab will be administered by IV infusion at a dose of 15 mg/kg on Day 1 of each 21-day cycle.
  Other Names: Avastin

SUMMARY:
This is a Phase IIIb, one arm, multicenter, open-label study primarily designed to evaluate the safety of atezolizumab + bevacizumab in participants with unresectable or unsuitable for locoregional treatments for metastatic HCC not previously treated with systemic therapy. As part of its secondary objectives, this study is also designed to evaluate the efficacy of atezolizumab and bevacizumab in these participants.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced or metastatic and/or unresectable HCC with diagnosis confirmed by histology or radiologically, following the AASLD criteria
* Disease that is not amenable to curative surgical and/or locoregional therapies, or progressive disease after surgical and /or locoregional therapies
* No prior systemic therapy (including systemic investigational agents) for HCC
* At least one measurable (per RECIST 1.1) untreated lesion detected by CT scan
* Patients who received prior local therapy such as radiofrequency ablation, percutaneous ethanol or acetic acid injection, cryoablation, high-intensity focused ultrasound, transarterial chemoembolization, transarterial embolization (excluding transarterial radioembolization.) are eligible provided the target lesion(s) have not been previously treated with local therapy or the target lesion(s) within the field of local therapy have subsequently progressed in accordance with RECIST version 1.1

Exclusion Criteria:

* Active or history of autoimmune disease or immune deficiency
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan
* Known fibrolamellar HCC, sarcomatoid HCC, or mixed cholangiocarcinoma and HCC
* Co-infection of HBV and HCV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-05-04 (Actual); Primary Completion 2024-04-26 (Actual); Study Completion 2024-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (25):
- Spain (25):
  - Hospital General Universitario de Elche, Elche, Alicante
  - Hospital Son Llatzer, Palma de Mallorca, Balearic Islands
  - Corporacio Sanitaria Parc Tauli, Sabadell, Barcelona
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital Provincial de Castellon, Castellon, Castellon
  - Complejo Hospitalario Universitario de Santiago (CHUS), Santiago de Compostela, LA Coruna
  - Hospital de Gran Canaria Dr. Negrin, Las Palmas de Gran Canaria, LAS Palmas
  - Hospital Universitario de Torrejon, Torrejón de Ardoz, Madrid
  - Clinica Universitaria de Navarra, Pamplona/iruña, Navarre
  - Hospital de Basurto, Bilbao, Vizcaya
  - Hospital General Univ. de Alicante, Alicante
  - Complejo Hospitalario Torrecardenas, Almería
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic i Provincial, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Complejo Hospitalario de Jaen-Hospital Universitario Medico Quirurgico, Jaén
  - Hospital Lucus Augusti, Lugo
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Clinica Universidad de Navarra Madrid, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Univ. Nuestra Señora de Valme, Seville
  - Hospital Universitari i Politecnic La Fe, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here ( https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 100 participants took part in the study in Spain from 04 May 2021 to 26 April 2024.
Pre-assignment Details: Participants with unresectable hepatocellular carcinoma (HCC) who received no prior systemic treatment and were considered unsuitable for locoregional therapy were enrolled in this study to receive a combination of atezolizumab plus bevacizumab until unacceptable toxicity or loss of clinical benefit.
Groups:
- Atezolizumab + Bevacizumab: Participants received atezolizumab, 1200 milligrams (mg), intravenously (IV), every 3 weeks (Q3W) along with bevacizumab, 15 milligrams per kilogram (mg/kg), IV, Q3W on Day 1 of each 21-day cycle until unacceptable toxicity or loss of clinical benefit.
Period: Overall Study
Arm/Group | Atezolizumab + Bevacizumab
Started | 100
Intent-to-treat Population (ITT) (ITT population included all screened participants (participants who signed the informed consent) who were eligible for the study.) | 99
Completed | 0
Not Completed | 100
Not completed — Progressive Disease | 2
Not completed — Physician Decision | 1
Not completed — Study Terminated by Sponsor | 31
Not completed — Withdrawal by Subject | 10
Not completed — Non-compliance With Study Drug | 1
Not completed — Lost to Follow-up | 4
Not completed — Death | 51

BASELINE CHARACTERISTICS:
Population: Safety population included all screened participants (participants who signed the informed consent) who received at least one full or partial dose of study treatment.
Groups:
- Atezolizumab + Bevacizumab: Participants received atezolizumab, 1200 mg, IV, Q3W along with bevacizumab, 15 mg/kg, IV, Q3W on Day 1 of each 21-day cycle until unacceptable toxicity or loss of clinical benefit.
Arm/Group | Atezolizumab + Bevacizumab
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.4 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 87
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27
  Not Hispanic or Latino | 73
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 99
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Discontinued Atezolizumab and/or Bevacizumab Due to Adverse Events (AE) of Grade ≥ 3
Description: AE is any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product, regardless of causal attribution. An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. The severity of AEs was assessed using National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0 (NCI CTCAE v5.0) with the following grades: Grade 1 = asymptomatic or mild symptoms; Grade 2 = minimal, local, or non-invasive intervention indicated; Grade 3 = severe or medically significant, but not immediately life-threatening; Grade 4 = life-threatening consequences or urgent intervention indicated and Grade 5 = death related to AE.
Time Frame: From Cycle 1 Day 1 up to 30 days after the final dose of the study drug or until initiation of another anti-cancer therapy, whichever occurred first (up to approximately 32 months)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Atezolizumab + Bevacizumab
Number analyzed (Participants) | 100
Participants | 19

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from initiation of study treatment to death from any cause. OS was analyzed using Kaplan-Meier (K-M) methods and Greenwood's formula. Any participant who did not die during the study was censored at the last known date to be alive.
Time Frame: Up to 35 months
Population: ITT population included all screened participants (participants who signed the informed consent) who were eligible for the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Atezolizumab + Bevacizumab
Number analyzed (Participants) | 99
months | 24.8 [18.55 to NA] — The upper limit of the 95% CI was not estimable due to insufficient number of participants with events.

3. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time from initiation of study treatment to the first occurrence of disease progression (PD) or death from any cause (whichever occurs first), as determined by the investigator according to Response Evaluation Criteria in Solid Tumours Version 1.1 (RECIST v1.1). PD was defined as at least a 20% increase in the sum of diameters (SOD) of target lesions, taking as reference the smallest SOD at prior timepoints (including baseline). In addition to the relative increase of 20%, the SOD must also demonstrate an absolute increase of ≥ 5 millimeters (mm). PFS was analyzed using K-M methods and Greenwood's formula. Any participant who did not experience disease progression or death during the study and were censored at the last known date to be alive or without disease progression.
Time Frame: Up to 35 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Atezolizumab + Bevacizumab
Number analyzed (Participants) | 99
months | 9.3 [7.01 to 12.40]

4. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR = percentage of participants with a complete or partial response (CR or PR), on 2 consecutive investigator assessments ≥ 4 weeks apart in participants with measurable disease at baseline as determined by the investigator according to RECIST v1.1. CR = disappearance of all target lesions and any pathological lymph nodes must have a reduction in short axis to < 10 mm. PR = at least a 30% decrease in the SOD of all target lesions, taking as reference the baseline SOD, in the absence of CR. Participants without a post-baseline tumor assessment were considered non-responders. 95% confidence interval (CI) was derived using Wilson score intervals. Percentages have been rounded off.
Time Frame: Up to 35 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Atezolizumab + Bevacizumab
Number analyzed (Participants) | 99
percentage of participants | 24.2 [16.9 to 33.5]

5. Secondary Outcome: Time to Progression (TTP)
Description: TTP was defined as the time from initiation of study treatment to the first occurrence of PD, as determined by the investigator according to RECIST v1.1. PD was defined as at least a 20% increase in the SOD of target lesions, taking as reference the smallest SOD at prior timepoints (including baseline). In addition to the relative increase of 20%, SOD must also demonstrate an absolute increase of ≥ 5 mm. TTP was analyzed using K-M methods and Greenwood's formula. Any participant who had no disease progression was censored at the last known date without disease progression.
Time Frame: Up to 35 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Atezolizumab + Bevacizumab
Number analyzed (Participants) | 99
months | 11.2 [8.30 to 13.59]

6. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the time from the first occurrence of a documented objective response (CR or PR) to PD or death from any cause (whichever occurs first), as determined by the investigator according to RECIST v1.1. CR was defined as disappearance of all target lesions and any pathological lymph nodes must have a reduction in short axis to < 10 mm. PR was defined as at least a 30% decrease in the SOD of all target lesions, taking as reference the baseline SOD, in the absence of CR. PD was defined as at least a 20% increase in the SOD of target lesions, taking as reference the smallest SOD at prior timepoints (including baseline). In addition to the relative increase of 20%, the SOD must also demonstrate an absolute increase of ≥ 5 mm. DOR was analyzed using K-M methods and Greenwood's formula. Any participant who did not experience disease progression or death during the study was censored at the last known date to be alive or without disease progression.
Time Frame: Up to 35 months
Population: ITT population included all screened participants (participants who signed the informed consent) who were eligible for the study. Overall number analyzed is the number of participants with an overall response of CR or PR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Atezolizumab + Bevacizumab
Number analyzed (Participants) | 24
months | 15.9 [7.87 to 23.74]

7. Secondary Outcome: Percentage of Participants Who Started Second-line Treatment
Description: Participants who started second-line of treatment were assessed. Percentages have been rounded off.
Time Frame: Up to 35 months
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Atezolizumab + Bevacizumab
Number analyzed (Participants) | 99
percentage of participants | 24.2

8. Secondary Outcome: Change From Baseline in International Normalized Ratio (INR)
Description: The INR is a standardized measure of the prothrombin time. Blood samples were collected from participants to evaluate coagulation parameters.
Time Frame: Baseline up to Cycle 42 (1 cycle = 21 days)
Population: Safety population included all screened participants (participants who signed the informed consent) who received at least one full or partial dose of study treatment. Overall number of participants analyzed is the number of participants with data available for analyses. Number analyzed is the number of participants with data available for analyses at the specified timepoints.
Measure: Mean (Standard Deviation); unit: INR of prothrombin time
Arm/Group | Atezolizumab + Bevacizumab
Number analyzed (Participants) | 99
INR of prothrombin time
  Baseline | 1.1 (0.1)
  Cycle 42: number analyzed (Participants) | 2
  Cycle 42 | 0.1 (0.0)

9. Secondary Outcome: Change From Baseline in Albumin-Bilirubin (ALBI) Score
Description: Blood samples were collected from participants to evaluate of ALBI grades. ALBI assessment grades of 1 to 3 was based on ALBI score calculation. ALBI score= log10 bilirubin (micromole per liter) [μmol/L] × 0.66 + albumin (grams per liter) [g/L] × -0.0852. ALBI score ≤ -2.60 = ALBI grade 1; -2.60 < ALBI score ≤ -1.39 = ALBI grade 2 and -1.39 < ALBI score = ALBI grade 3.
Time Frame: Baseline up to Cycle 42 (1 cycle = 21 days)
Population: Safety population included all screened participants (participants who signed the informed consent) who received at least one full or partial dose of study treatment. Number analyzed is the number of participants with data available for analyses at the specified timepoints.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Atezolizumab + Bevacizumab
Number analyzed (Participants) | 100
score
  Baseline | -2.7 (0.4)
  Cycle 42: number analyzed (Participants) | 2
  Cycle 42 | 0.4 (0.4)

10. Secondary Outcome: Percentage of Participants With Ascites and/or Hepatic Encephalopathy
Description: Deterioration of hepatic function was monitored by presence of ascites and/or hepatic encephalopathy.
Time Frame: Up to approximately 32 months
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Atezolizumab + Bevacizumab
Number analyzed (Participants) | 100
percentage of participants | 17

ADVERSE EVENTS:
Time Frame: AEs and SAEs: From Cycle 1 Day 1 up to 30 days after the final dose of the study drug or until initiation of another anti-cancer therapy, whichever occurred first (up to approximately 32 months). All cause mortality: Up to 35 months
Description: Safety population included all screened participants (participants who signed the informed consent) who received at least one full or partial dose of study treatment.
Groups:
- Atezolizumab + Bevacizumab:: Participants received atezolizumab, 1200 mg, IV, Q3W along with bevacizumab, 15 mg/kg, IV, Q3W on Day 1 of each 21-day cycle until unacceptable toxicity or loss of clinical benefit.
Arm/Group | Atezolizumab + Bevacizumab:
All-Cause Mortality (participants affected / at risk) | 51/100
Serious Adverse Events (participants affected / at risk) | 46/100
Other Adverse Events (participants affected / at risk) | 98/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atezolizumab + Bevacizumab: (N=100)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 2 (2)
Hepatic Function Abnormal (Hepatobiliary disorders) | 1 (1)
Immune-Mediated Hypothyroidism (Endocrine disorders) | 1 (1)
Pyrexia (General disorders) | 2 (2)
Tumour Associated Fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Duodenal Ulcer Haemorrhage (Gastrointestinal disorders) | 1 (1)
Gastric Perforation (Gastrointestinal disorders) | 1 (1)
Intestinal Perforation (Gastrointestinal disorders) | 1 (1)
Intra-Abdominal Haemorrhage (Gastrointestinal disorders) | 1 (1)
Oesophageal Varices Haemorrhage (Gastrointestinal disorders) | 3 (3)
Hepatic Enzyme Increased (Investigations) | 1 (2)
Myelin Oligodendrocyte Glycoprotein Antibody-Associated Disease (Nervous system disorders) | 1 (1)
Tubulointerstitial Nephritis (Renal and urinary disorders) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 3 (3)
Abdominal Pain (Gastrointestinal disorders) | 2 (2)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 2 (2)
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 2 (2)
Haemoperitoneum (Gastrointestinal disorders) | 1 (1)
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 1 (1)
Intestinal Obstruction (Gastrointestinal disorders) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Pneumonia Pneumococcal (Infections and infestations) | 2 (2)
Urinary Tract Infection (Infections and infestations) | 2 (2)
Abdominal Sepsis (Infections and infestations) | 1 (1)
Biliary Sepsis (Infections and infestations) | 1 (1)
Covid-19 (Infections and infestations) | 1 (1)
Covid-19 Pneumonia (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (2)
Infective Exacerbation Of Chronic Obstructive Airways Disease (Infections and infestations) | 1 (1)
Peritonsillar Abscess (Infections and infestations) | 1 (1)
Pneumonia Aspiration (Infections and infestations) | 1 (1)
Respiratory Tract Infection (Infections and infestations) | 1 (1)
Spontaneous Bacterial Peritonitis (Infections and infestations) | 1 (1)
Hepatic Encephalopathy (Nervous system disorders) | 5 (5)
Spinal Cord Compression (Nervous system disorders) | 2 (2)
Encephalopathy (Nervous system disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
General Physical Health Deterioration (General disorders) | 2 (2)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hip Fracture (Injury, poisoning and procedural complications) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Tibia Fracture (Injury, poisoning and procedural complications) | 1 (1)
Wound Dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Wound Evisceration (Injury, poisoning and procedural complications) | 1 (1)
Cholecystitis Acute (Hepatobiliary disorders) | 1 (1)
Jaundice (Hepatobiliary disorders) | 1 (1)
Blood Bilirubin Increased (Investigations) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 1 (1)
Oesophageal Variceal Ligation (Surgical and medical procedures) | 1 (1)
Spinal Laminectomy (Surgical and medical procedures) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Confusional State (Psychiatric disorders) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 1 (1)
Peripheral Ischaemia (Vascular disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Subdiaphragmatic Abscess (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atezolizumab + Bevacizumab: (N=100)
Diarrhoea (Gastrointestinal disorders) | 30 (64)
Abdominal Pain (Gastrointestinal disorders) | 22 (32)
Constipation (Gastrointestinal disorders) | 20 (22)
Vomiting (Gastrointestinal disorders) | 13 (15)
Abdominal Pain Upper (Gastrointestinal disorders) | 11 (13)
Nausea (Gastrointestinal disorders) | 11 (17)
Ascites (Gastrointestinal disorders) | 9 (11)
Dry Mouth (Gastrointestinal disorders) | 6 (8)
Dyspepsia (Gastrointestinal disorders) | 6 (7)
Haemorrhoids (Gastrointestinal disorders) | 5 (5)
Asthenia (General disorders) | 46 (78)
Pyrexia (General disorders) | 13 (16)
Oedema Peripheral (General disorders) | 11 (16)
Mucosal Inflammation (General disorders) | 9 (14)
Pain (General disorders) | 7 (8)
Fatigue (General disorders) | 5 (6)
Oedema (General disorders) | 5 (5)
Covid-19 (Infections and infestations) | 21 (22)
Nasopharyngitis (Infections and infestations) | 12 (13)
Respiratory Tract Infection (Infections and infestations) | 7 (8)
Back Pain (Musculoskeletal and connective tissue disorders) | 14 (17)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 (19)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 7 (8)
Hypertension (Vascular disorders) | 42 (56)
Pruritus (Skin and subcutaneous tissue disorders) | 24 (29)
Rash (Skin and subcutaneous tissue disorders) | 5 (7)
Skin Lesion (Skin and subcutaneous tissue disorders) | 5 (5)
Blood Bilirubin Increased (Investigations) | 9 (10)
Lipase Increased (Investigations) | 9 (14)
Platelet Count Decreased (Investigations) | 9 (9)
Amylase Increased (Investigations) | 6 (8)
Weight Decreased (Investigations) | 6 (6)
Alanine Aminotransferase Increased (Investigations) | 5 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (11)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Headache (Nervous system disorders) | 13 (15)
Dysgeusia (Nervous system disorders) | 5 (5)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 9 (10)
Hyperbilirubinaemia (Hepatobiliary disorders) | 10 (13)
Hypertransaminasaemia (Hepatobiliary disorders) | 8 (10)
Proteinuria (Renal and urinary disorders) | 18 (23)
Thrombocytopenia (Blood and lymphatic system disorders) | 11 (18)
Anaemia (Blood and lymphatic system disorders) | 6 (8)
Hypothyroidism (Endocrine disorders) | 14 (14)
Insomnia (Psychiatric disorders) | 10 (11)
Decreased Appetite (Metabolism and nutrition disorders) | 22 (31)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigators are free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2023-03-16): https://cdn.clinicaltrials.gov/large-docs/86/NCT04732286/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-26): https://cdn.clinicaltrials.gov/large-docs/86/NCT04732286/SAP_001.pdf